CLINICAL TRIAL: NCT04498481
Title: TREATMENT AND MONITORING PATTERNS AND CLINICAL OUTCOMES IN PATIENTS RECEIVING PALBOCICLIB PLUS AROMATASE INHIBITOR OR PALBOCICLIB PLUS FULVESTRANT AS TREATMENT OF HORMONE RECEPTOR POSITIVE (HR+)/HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR 2 NEGATIVE (HER2-) ADVANCED OR METASTATIC BREAST CANCER IN A REAL WORLD COMMUNITY ONCOLOGY SETTING
Brief Title: TREATMENT AND MONITORING PATTERNS AND CLINICAL OUTCOMES IN PATIENTS RECEIVING PALBOCICLIB COMBINATION TREATMENT (WITH AI OR FULVESTRANT) FOR HR+/HER2- A/MBC IN A COMMUNITY ONCOLOGY SETTING.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481095
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast cancer patients: HR+/HER2- advanced/metastatic breast cancer patients in the USA.

SUMMARY:
This is a retrospective, observational study that will document the treatment and monitoring patterns and clinical outcomes of patients diagnosed with HR+/HER2- a/mBC who received Palbociclib combination therapy with aromatase inhibitors or fulvestrant in the a/mBC community oncology setting.

ELIGIBILITY:
Inclusion Criteria:

Patients who are represented in the Vector Oncology Data Warehouse who meet all of the following criteria will be eligible for inclusion in the study.

* Female.
* Diagnosis of female breast cancer with evidence of metastatic disease or advanced disease.
* Diagnosis (confirmed by clinical review) of advanced or metastatic breast cancer at any time, defined as breast cancer at stage IIIb, stage IIIc, or stage IV or identified as having distant metastasis.
* Indication in the record of ER or PR positive disease, or absence of any indication of ER and PR negative disease (ie, patients are eligible without affirmative indication of ER/PR+ status as long as ER/PR- indication is not present).
* Receipt of a palbociclib plus aromatase inhibitor (AI) or palbociclib plus fulvestrant regimen on 2/3/2015 or later in the advanced and metastatic setting. Data collection will prioritize accrual of patients with 1L use of palbociclib plus AI and with 2L use of palbociclib plus fulvestrant before collecting other use of palbociclib users.
* Age greater than or equal to 18 years at A/MBC diagnosis.

Exclusion Criteria:

-There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will include adult patients aged 18 years and older, diagnosed with HR+/HER2- a/mBC who received Palbociclib combination therapy with AI or fulvestrant on or after 2/3/2015.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving various cancer treatment regimens | A/MBC diagnosis through end of study (assessed up to 24 months)
Proportion of patients receiving each therapy sequence across lines | A/MBC diagnosis through end of study (assessed up to 24 months)
Treatment persistence | A/MBC diagnosis through end of study (assessed up to 24 months)
Progression Free Survival (PFS) | A/MBC diagnosis through end of study (assessed up to 24 months)
Overall Survival (OS) | A/MBC diagnosis through end of study (assessed up to 24 months)
Tumor response rate | A/MBC diagnosis through end of study (assessed up to 24 months)
Proportion of patients that experience dose adjustment | A/MBC diagnosis through end of study (assessed up to 24 months)
Proportion of patients who discontinue therapy | A/MBC diagnosis through end of study (assessed up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer United States, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Robert N, Chen C, Doan J, Venkatasetty D, Espirito JL, Aguilar KM. Real-world study of patients with HR+/ HER2- metastatic breast cancer treated with palbociclib and fulvestrant. Future Oncol. 2025 Jan;21(1):83-94. doi: 10.1080/14796694.2024.2442302. Epub 2025 Jan 15. PMID 39810652
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481095